CLINICAL TRIAL: NCT00004075
Title: A Phase I Trial of 17-Allylaminogeldanamycin (17-AAG) in Solid Tumor and Lymphoma Patients
Brief Title: 17-N-Allylamino-17-Demethoxygeldanamycin in Treating Patients With Solid Tumors That Cannot Be Removed By Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Charles Erlichman, M.D., Mayo Clinic Cancer Center
Purpose: Treatment
Other Study IDs: CDR0000067283; U01CA069912 (NIH); P30CA015083 (NIH); 990102 (Other: Mayo Clinic Cancer Center)
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-08

CONDITIONS: Lymphoma; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent mycosis fungoides/Sezary syndrome; recurrent adult grade III lymphomatoid granulomatosis; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — tanespimycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: tanespimycin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase I trial is studying the side effects and best dose of 17-N-allylamino-17-demethoxygeldanamycin in treating patients with solid tumors that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose and dose-limiting toxicity of 17-N-allylamino-17-demethoxygeldanamycin (17-AAG), administered at 2 different dosing schedules, in patients with unresectable solid tumors.
* Determine the pharmacokinetics of this drug in these patients.
* Assess the effect of this drug on heat shock protein chaperone complex components and client proteins in lymphoma tissue obtained pre- and post-treatment in patients with relapsed lymphoma.
* Determine any response to this drug in these patients.

OUTLINE: This is a dose-escalation study. Patients are assigned to 1 of 2 treatment groups.

* Group I: Patients receive 17-N-allylamino-17-demethoxygeldanamycin (17-AAG) IV over 1 hour on days 1, 8, and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
* Group II: Patients receive 17-AAG IV over 1 hour on days 1, 4, 8, and 11. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Cohorts of 1-6 solid tumor patients receive escalating doses of 17-AAG until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose-limiting toxicity.

Once the MTD is determined, 10 patients with either lymphoma or superficial solid tumors accessible for biopsy are treated as in group II at the MTD.

Patients are followed for 3 months.

PROJECTED ACCRUAL: A total of 58-130 patients (30-72 for group I and 28-58 for group II) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* One of the following diagnoses:

  * Histologically or cytologically confirmed solid tumor*

    * Unresectable disease
  * Hodgkin's or non-Hodgkin's lymphoma

    * Relapsed disease
    * Failed at least 1 prior therapy
    * Neoplastic cells are accessible through biopsy NOTE: *Only patients with biopsy-accessible superficial tumors or lymphoma are eligible once the maximum tolerated dose has been determined
* No known standard therapy that is potentially curative or definitely capable of extending life expectancy exists
* No CNS metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST no greater than 2.5 times ULN
* Alkaline phosphatase no greater than 2 times ULN (5 times ULN if liver involvement)

Renal:

* Creatinine no greater than 1.25 times ULN OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective nonhormonal contraception
* No uncontrolled infection
* No seizure disorder
* No history of serious allergic reaction to eggs

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* More than 4 weeks since prior immunotherapy
* More than 4 weeks since prior biologic therapy
* No concurrent immunotherapy
* No concurrent routine or prophylactic use of a colony-stimulating factor (e.g., filgrastim [G-CSF] or sargramostim [GM-CSF])

Chemotherapy:

* More than 4 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas) and recovered from acute and reversible toxic effects
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent birth control pills
* No concurrent steroids as anti-emetics

Radiotherapy:

* More than 4 weeks since prior radiotherapy
* No prior radiotherapy to more than 25% of the bone marrow
* No prior radiopharmaceuticals
* No concurrent radiotherapy

Surgery:

* Not specified

Other:

* No concurrent 3A4 enzyme inhibitors (e.g., verapamil, erythromycin, miconazole, or ketoconazole)
* No concurrent investigational ancillary therapy
* No concurrent enrollment in another study involving a pharmacologic agent (e.g., drugs, biologics, immunotherapy approaches, or gene therapy) for symptom control or therapeutic intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-08; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Erlichman, MD, Study Chair — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States